CLINICAL TRIAL: NCT06621199
Title: A Prospective, Single-arm, Multi-center, Phase 2 Clinical Study of Mitoxantrone Hydrochloride Liposome in Combination With Cytarabine and Venetoclax Regimen in Newly Diagnosed Elderly AML
Brief Title: Mitoxantrone Hydrochloride Liposome in Combination With Cytarabine and Venetoclax Regimen in Newly Diagnosed Elderly AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-AML-K15
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified MAV regimen (Experimental): Mitoxantrone hydrochloride liposome ×1 day, cytarabine × 5 days combined with venetoclax as induction regimen
  Interventions: Drug: Mitoxantrone hydrochloride liposome; Drug: Cytarabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride liposome — Mitoxantrone hydrochloride liposome 24 mg/m^2 on day 1, every 4 weeks
Drug: Cytarabine — Cytarabine 100 mg/m^2 on day 1-5, every 4 weeks
Drug: Venetoclax — Venetoclax 100 mg on day 2，200 mg on day 3，400 mg on day 4-10, every 4 weeks

SUMMARY:
This is a phase 2 study to evaluate the efficacy and safety of mitoxantrone hydrochloride liposome in combination with cytarabine and venetoclax (MAV) regimen in newly diagnosed elderly AML. To account, conservatively, for a 10% dropout rate before study completion, we planned to include 42 patients. The primary endpoint is 2-year event free survival(EFS).

DETAILED DESCRIPTION:
The optimal induction chemotherapy regimen for newly diagnosed elderly AML patients who are eligible for intense chemotherapy is currently not well defined. Mitoxantrone hydrochloride liposome (Lipo-MIT) is an innovative anthracycline nano-drug, which has been demonstrated favorable pharmacokinetic characteristics, high cardiac safety, and shown preliminary efficacy in adult AML. Thus, we designed a prospective, single-arm, phase 2 trial to explore the efficacy and safety of Lipo-MIT in combination with cytarabine and venetoclax (MAV) regimen in newly diagnosed elderly AML.

The induction therapy is a combination of Lipo-MIT (24 mg/m^2, day 1), cytarabine(100mg/m^2, day 1-5) and venetoclax (200mg day 2, 300mg day 3, 400mg day 4-10,), and would be applied for two cycles. Patients who achieve CR/CRi after using MAV induction regimen will receive the consolidation therapy according to the patients' cytogenetic-molecular risk stratification and maintenance therapy. After completion of the treatment phase, patients entered the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.
2. Aged 60-70 years (including boundary values 60 and 70);
3. Newly diagnosed primary AML according to the WHO 2022 classification.
4. Physical status score of Eastern Oncology Collaboration Group (ECOG) : 0-2.
5. Life expectancy ≥ 3 months.
6. ALT/AST≤2.5 ULN (for subjects with hepatic infiltration≤5 ULN); Total bilirubin≤1.5 ULN (for subjects with hepatic infiltration≤3 ULN); Serum creatinine≤1.5 ULN.

Exclusion Criteria:

1. Subjects meet any of the following conditions:

   1. Acute promyelocytic leukemia;
   2. Secondary AML caused by chemotherapy and/or radiotherapy to treat solid tumor or antecedent hematological disorders such as MDS, MPN, MDS/MPN;
   3. AML following blast transformation of prior chronic myeloid leukemia;
   4. Central nervous system (CNS) leukemia;
2. Subjects with malignant tumors (excluding cured skin basal cell carcinoma, cervical carcinoma in situ, and other malignant tumors that have not been treated and effectively controlled within the past 5 years) within the past 5 years.
3. Subjects who have received anthracycline pretreatment or other anti-AML treatments (except for hydroxyurea, leukapheresis and other leukocyte-lowering treatments);
4. Subjects who received strong or moderate CYP3A inducers/inhibitors or P-glycoprotein (P-gp) inhibitors within 7 days before starting study treatment;
5. Subjects who are unable to take oral medications or have malabsorption syndrome;
6. Cardiac function and disease conform to one of the following conditions:

   1. Long QTc syndrome or QTc interval >480 ms;
   2. Complete left bundle branch block, degree II or III atrioventricular block;
   3. Severe, uncontrolled arrhythmia requiring medical treatment;
   4. New York Heart Association(NYHA) classification ≥ grade II;
   5. Cardiac ejection fraction (EF) was less than 50%;
   6. A history of myocardial infarction, unstable angina pectoris, severely unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically severe pericardial disease, or electrocardiogram evidence of acute ischemic or active conduction abnormalities within 6 months prior to enrollment;
7. Uncontrolled systemic diseases (such as advanced infections, uncontrolled hypertension, diabetes, etc.);
8. Human immunodeficiency virus (HIV) infection (HIV antibody positive);
9. HBsAg or HBcAb positive, with HBV-DNA≥1x10^3 copies/mL; HCV Ab positive, with HCV-RNA≥1x10^3 copies/mL;
10. A history of immediate or delayed allergy to similar drug and excipients of the investigate drug.
11. With a history of severe neurological or psychiatric illness.
12. Not suitable for this study as decided by the investigator.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year event-free survival (EFS) rate | up to 2 years
  Defined for all patients in the study. Measured from day 1 of treatment to the date of treatment failure, hematologic relapse from CR/CRi or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Composite complete remission (CRc) rate of induction therapy | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  Complete remission plus complete remission with incomplete hematologic recovery (CR+CRi). Response is assessed according to the the European LeukemiaNet (ELN) 2022 criteria.
Overall response rate (ORR) of induction therapy | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  CR+CRi+morphologic leukemia-free state+partial remission (CR+CRi+MLFS+PR). Response is assessed according to the the European LeukemiaNet (ELN) 2022 criteria.
Relapsed-free survival (RFS) | up to 2 years
  Defined only for patients achieving CR or CRi. Measured from the date of achievement of remission until the date of hematologic relapse or death from any cause.
Overall survival (OS) | up to 2 years
  Defined for all patients in the study. Measured from day 1 of treatment to the date of death from any cause.
Rate of CR/CRi without measurable residual disease after induction therapy | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  Percentage of participants who achieve a CR MRD-/CRi MRD- as defined by investigators based on ELN 2022 criteria. MRD level is detected by flow cytometry and negtive MRD is defined as MRD value <0.1%.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From day 1 of treatment to 28 days after the last dose
  The safety of the regimen was evaluated by NCI-CTC AE 5.0 standard which including hematologic and non-hematologic toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China